CLINICAL TRIAL: NCT07129655
Title: Cholangitis Definition and Treatment After Kasai Hepatoportoenterostomy for Biliary Atresia: a Feasibility Study
Brief Title: Cholangitis Definition and Treatment After Kasai Hepatoportoenterostomy for Biliary Atresia: TRACK-BA Study (TRacking Cholangitis Post Kasai in Biliary Atresia)
Acronym: TRACK-BA
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Calinescu Ana M., PD Dr Ana M. Calinescu, University Hospital, Geneva
Other Study IDs: 2021-01251
Record Dates: First submitted 2025-08-11; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Biliary Atresia, Kasai Portoenterostomy Status; Cholangitis
Keywords: biliary atresia; Kasai hepatoportoenterostomy; acute cholangitis
MeSH Terms: conditions — Biliary Atresia; Cholangitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A sample size of 40 patients is targeted, with 20 in each group (suspected and confirmed).: Patients with a suspected diagnosis cholangitis within 1 year after Kasai hepatoportoenterostomy:
  This includes patients for whom
  1. cholangitis will not be finally confirmed ,
  2. cholangitis is finally confirmed.

SUMMARY:
Biliary atresia is a rare liver disease affecting newborns. In those babies bile ducts are blocked, and bile cannot flow from the liver to the intestines. Biliary atresia patients require a special surgery called "Kasai operation" to restore the bile flow. A common and serious problem after surgery is an infection of the bile ducts, called cholangitis, which can damage the liver and lead an earlier need for liver transplantation.

In 2022, a group of international experts led by the Swiss Pediatric Liver Center from the HUG created new guidelines to help identify and treat cholangitis more consistently.

This study will test how well these new definitions work in real life of hospitals. Over one year, physicians will collect data on children in whom they suspect cholangitis in the first year after their Kasai. The goal is to see whether these new definitions are applicable in the clinical setting.

The study will involve around 40 patients and will use secure methods to store data. The findings will help improve how cholangitis is diagnosed and treated, making care more effective and consistent for children with biliary atresia.

DETAILED DESCRIPTION:
This prospective, observational study will be conducted across hospitals managing pediatric biliary atresia patients. Data on suspected cholangitis cases in the first year post Kasai hepatoportoenterostomy will be collected by mini-teams of three healthcare providers over twelve months. Data will be anonymized, and the study will adhere to international ethical standards.

Inclusion Criteria:

* Patients with biliary atresia suspected of cholangitis within one year post Kasai hepatoportoenterostomy.
* Data from specialties including pediatric surgery, pediatric hepatology, and pediatric emergency care.

Exclusion Criteria:

• Recurrent cholangitis or cholangitis after one-year post Kasai hepatoportoenterostomy.

Definitions: Cholangitis will be defined by clinical confirmation, improvement with antimicrobial therapy, and lab value changes.

Primary Aim: To assess the application of consensus definitions for suspected and confirmed cholangitis.

Secondary Aim: To evaluate the proposed duration of treatment for cholangitis and compare it to clinical practice.

Data Collection: Data will be stored using the secure REDCap platform, managed by the University of Geneva. Local investigators are responsible for ethical approvals.

Expected Results: This study will assess the practicality of applying expert panel definitions for cholangitis after Kasai hepatoportoenterostomy and gather feedback from clinicians. A sample size of 40 patients is targeted, with 20 in each group (suspected and confirmed). Findings will help refine diagnostic criteria.

ELIGIBILITY:
Inclusion Criteria:

* patients with a suspected diagnosis cholangitis within 1 year after Kasai hepatoportoenterostomy

Exclusion Criteria:

* recurrent cholangitis, cholangitis >1 year after Kasai

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Definition and treatment of cholangitis after Kasai hepatoportoenterostomy were established after an international consensus of a panel of experts led by the Swiss Pediatric Liver Center within the Geneva University Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
To assess the applicability of the definitions for suspected and confirmed cholangitis. | 12 months

SECONDARY OUTCOMES:
Duration of treatment for suspected and confirmed cholangitis | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The Individual Participant Data (IPD) to be shared will include anonymised clinical, demographic, and outcome data relevant to the study objectives.
  Demographic data: Age, sex, weight, gestational age at birth. Clinical data: Diagnosis date, baseline lab values, imaging results. Treatment data: Assigned group, medications used, dates of intervention. Follow-up data: Lab results over time, response to treatment.
Supporting Information: Study Protocol, SAP, Analytic Code
Access Criteria: There will be three physicians responsible per site, as well as one dedicated person in charge of data entry into the database.

REFERENCES:
- [Background] Madadi-Sanjani O, Calinescu AM, Rock N, McLin VA, Uecker M, Kuebler JF, Petersen C, Wildhaber BE. Retrospective analysis of the standardized BARD criteria for acute cholangitis in biliary atresia patients. JPGN Rep. 2024 Apr 12;5(3):309-316. doi: 10.1002/jpr3.12071. eCollection 2024 Aug. PMID 39149194
- [Background] Calinescu AM, Madadi-Sanjani O, Mack C, Schreiber RA, Superina R, Kelly D, Petersen C, Wildhaber BE. Cholangitis Definition and Treatment after Kasai Hepatoportoenterostomy for Biliary Atresia: A Delphi Process and International Expert Panel. J Clin Med. 2022 Jan 19;11(3):494. doi: 10.3390/jcm11030494. PMID 35159946

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study protocol and statistical analysis plan (2025-04-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT07129655/Prot_SAP_000.pdf
  • Study Protocol: Case Report Form (2025-04-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT07129655/Prot_001.pdf